CLINICAL TRIAL: NCT02310880
Title: Efficacy of Enhancing Low Vision Mobility Thru Visual Training in Virtual World
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: X100716003
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-12

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low vision (virtual street training): Low vision subjects trained in virtual streets and observed in real streets
- Low vision (real street training): Low vision subjects trained in real streets and observed in real streets

SUMMARY:
Low vision patients have difficulty acquiring sufficient visual information in a timely manner for the purpose of performing challenging daily tasks, such as traveling independently and safely through busy streets. The advance of virtual reality techniques has provided a potential platform for training low vision patients to use their remaining vision more efficiently, but the key issue is always whether the patient's visual experiences in a virtual world can be transferred to the real world. The proposed study is designed to provide definite answer to this question.

DETAILED DESCRIPTION:
NEI's National Plan for Eye and Vision Research has identified Low Vision and Blindness Rehabilitation as one of the most pressing needs and opportunities in vision research. Since most low vision (LV) patients nowadays have useable vision, an important aspect of LV rehabilitation is to maximize the use of the patient's remaining vision. Visual skills are especially important in tasks such as traveling independently through busy streets, in which distant, rapidly changing events have direct impact on the patient's task efficiency and safety. The patient has to learn new information acquisition skills to compensate for their impaired vision. Current LV training for such skills is done on real streets in a one-on-one, trainer/trainee sessions. This way of training, however, usually does not expose clients to all the circumstances that they need to deal with, usually does not provide graded levels of task difficulty and repeatable conditions that facilitate learning, and cannot meet the needs of the majority of LV patients because of the shortage and the high cost of LV trainers. The advances of virtual reality (VR) technology have made it possible and affordable to realistically simulate complex and dynamic visual and auditory environments to facilitate LV rehabilitation. However, the most important first step in applying VR technologies to LV rehabilitation is to determine whether the visual experiences of a LV person can be transferred to the real world. Only when a positive transfer of visual skills is confirmed, can subsequent development of comprehensive VR training systems for all aspects of LV rehabilitation become worthwhile. The purpose of this study is to accomplish this first step. A set of visual skills for a most visually challenging task, crossing a signal-controlled street, is selected from standard orientation and mobility curriculum to study virtual experience transfer. Existing technology are used to build a desktop computer-based VR simulator that can generate virtual street intersection scenarios that contain visual and auditory information required for practicing the skills to be studied. Computer generated street intersections with pedestrians, traffic and control signals are projected to a large screen for the participant to view, like a movie. Twenty LV persons are recruited from a university LV rehabilitation facility. They are randomly assigned to practicing the selected visual skills at real or virtual street intersections. Their skill levels are evaluated at real intersections before and immediately after their scheduled training. The primary outcome of interest is the mean change of visual skills between pre- and post-training evaluations in the two groups. The training is not a rehabilitation intervention because only the changes in visual/audio information gathering skills are trained and observed. The participants are trained and evaluated on the sidewalks of the real and virtual street. They are never allowed to step down the curb to avoid exposure to any danger. The long-term goal is to develop interactive VR training systems that have multiple sensory and motor input and output modules and that incorporate the collective experiences of the LV rehabilitation profession. Adding such systems to LV curriculum can greatly improve the affordability, accessibility, efficiency and the scope of LV rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory and have independent traveling as one of their rehabilitation goals.
* Participants with central field loss should have best corrected binocular visual acuity between 20/200 and 20/1000, but with relatively intact peripheral visual field (>80o).
* Participants with peripheral visual field loss should have >20/63 visual acuity and no more than 20 deg diameter but not less than 8 deg diameter visual field in the better eye.

Exclusion Criteria:

* Participants who have a mixture of central and peripheral field loss.
* Previous or current recipient of O&M training.
* Participants who have plans to receive O&M training during the study period.
* Age younger than 19 or older than 81.
* Significant cognitive impairment as determined with the Short Portable Mental Status Questionnaire (≥2 errors); inability to understand and speak English.
* Severe hearing impairment that interferes with interactions with O&M specialists.
* Inability or unwillingness to make visits required by the study.
* Not living in the Birmingham-Jefferson county area.
* Persons who have a history of epilepsy or who are prone to motion sickness or simulator aftereffect, determined by an epileptic seizure history inquiry and a Motion Sickness History Questionnaire.

Ages: 19 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low vision participants will be recruited from the patient populations of the Clinics of UAB School of Optometry and UAB Center for Low Vision Rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The percentage of dangerous street crossing decisions and the street crossing decision safety scores | 3-5 1-hour visits
  The percentage of dangerous street crossing decisions is determined at real street corners during pre- and post-training evaluation sessions. The subject is asked to say "GO" when she feels it is the safest time to cross the street. A crossing decision is scored as dangerous if it is initiated in the red traffic light cycle or if there is < 25% of the "WALK" cycle left. The percentage is the total number of dangerous decisions divided by the total number of crossing decisions made during one evaluation session. The safety of a crossing decision is further quantified by recording the decision timing using a stopwatch and by converting the recorded time to a safety score. The safety score is a continuous scale between 0 and 1.0. The larger the safety score, the safer is the crossing decision. A statistically significant reduction in the percentage dangerous crossing decisions and an increase in the safety scores after training is an indication of successful skill learning and transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Clinical Eye Research Facility, Birmingham, Alabama, United States